CLINICAL TRIAL: NCT04691648
Title: An Observational Study to Assess the Safety of Xospata® 40 mg Tablet When Administered in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML) With FMS-Like Tyrosine Kinase 3 (FLT3) Mutation
Brief Title: A Study to Assess the Safety of Xospata in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML) With FMS-Like Tyrosine Kinase 3 (FLT3) Mutation
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 2215-PV-001
Record Dates: First submitted 2020-12-30; First posted 2020-12-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia With FMS-like Tyrosine Kinase (FLT3) Mutation
Keywords: Gilteritinib; Xospata; Relapsed or refractory Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute | interventions — gilteritinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Xospata: Patients who receive Xospata® 40 mg tablet in routine clinical practice according to the drug label approved at the time of marketing authorization.
  Interventions: Drug: Gilteritinib Exposure

INTERVENTIONS:
Drug: Gilteritinib Exposure — Oral
  Other Names: Xospata

SUMMARY:
The objective of this study is to describe the observed safety profile of Xospata® 40 mg tablet when administered in patients with relapsed or refractory AML with FLT3 mutation in routine clinical practice in Korea.

DETAILED DESCRIPTION:
This study is being mandated by Ministry of Food and Drug Safety (MFDS) as a part of the Korea-Risk Management Plan (K-RMP) to assess safety in patients with relapsed or refractory AML with FLT3 mutation in routine clinical practice in Korea. This study collects data for 54 months according to the purpose of this study in routine clinical practice as an observational study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive Xospata® 40 mg tablet according to the drug label approved at the time of marketing authorization in routine clinical practice.
* Patients who voluntarily signed the written informed consent form.

Exclusion Criteria:

* Patients who meet the section 'Do not administer to the following patients' in the precautions for use given at the time of marketing authorization.
* Patients who use the drug for an off-label purpose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving Xospata® 40 mg tablet according to the drug label for 54 months from the start date of marketing in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2025-05-04 (Actual); Study Completion 2025-05-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Drug Reactions (ADRs) related to important identified and/or potential risks | Up to a maximum of 54 months (until 30 days after the last dose)
  An Adverse Drug Reaction refers to any unfavorable and unintended reaction occurring with a normal administration or use of the medicinal product that a causal relationship to the medicinal product cannot be ruled out. Number of ADRs related to important identified risks such as posterior reversible encephalopathy syndrome (PRES), QT prolongation, differentiation syndrome, and/or important potential risks such as pancreatitis, embryo-fetal lethality, suppressed fetal growth and teratogenicity, will be recorded.
Number of participants with serious ADRs related to important identified and/or potential risks | Up to a maximum of 54 months (until 30 days after the last dose)
  An ADR refers to any unfavorable and unintended reaction occurring with a normal administration or use of the medicinal product that a causal relationship to the medicinal product cannot be ruled out. Number of ADRs related to important identified risks such as posterior reversible encephalopathy syndrome (PRES), QT prolongation, differentiation syndrome, and/or important potential risks such as pancreatitis, embryo-fetal lethality, suppressed fetal growth and teratogenicity, will be recorded. An ADR is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes: results in death, is life-threatening, results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, results in congenital anomaly or birth defect, requires inpatient hospitalization or prolongation of hospitalization, or other medically important event.

SECONDARY OUTCOMES:
Number of participants with ADRs related to identified risks and considered not important | Up to a maximum of 54 months (until 30 days after the last dose)
  An ADR refers to any unfavorable and unintended reaction occurring with a normal administration or use of the medicinal product that a causal relationship to the medicinal product cannot be ruled out. Number of ADRs related to identified risks but considered not important, such as other ADRs described by the Korean package insert, will be recorded. An ADR is considered "serious" if, in the view of either the investigator or Sponsor, it results in any of the following outcomes: results in death, is life-threatening, results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, results in congenital anomaly or birth defect, requires inpatient hospitalization or prolongation of hospitalization, or other medically important event.
Number of participants with AEs | Up to a maximum of 54 months (until 30 days after the last dose)
  An AE is defined as any untoward medical occurrence in a subject administered a study drug, and which does not necessarily have to have a causal relationship with this treatment. An AE is considered "serious" if, in the view of either the investigator or Sponsor, it results in any of the following outcomes: results in death, is life-threatening, results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, results in congenital anomaly or birth defect, requires inpatient hospitalization or prolongation of hospitalization, or other medically important event. Causal relationship between the study drug is judged by medically qualified investigator either as certain, probable/likely, possible, unlikely, conditional/unclassified or unassessable/unclassifiable.

CONTACTS AND LOCATIONS:
Overall Officials: Astellas Pharma Korea, Inc., Study Director — Astellas Pharma Korea, Inc.
Locations (10):
- South Korea (10):
  - Site KR82013, Wŏnju, Gangwon-do
  - Site KR82006, Goyang-si, Gyeonggi-do
  - Site KR82003, Jeollanam-do, Hwasun-gun
  - Site KR82011, Busan
  - Site KR82010, Daegu
  - Site KR82001, Incheon
  - Site KR82004, Seoul
  - Site KR82005, Seoul
  - Site KR82009, Seoul
  - Site KR82007, Seoul

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.